CLINICAL TRIAL: NCT06395961
Title: Effect of New High Ankle Block on Wound Healing After the Operation of Debridement of Diabetes Foot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XuzhouCH-WK1
Record Dates: First submitted 2024-02-27; First posted 2024-05-02 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Wound Heal; Diabetic Foot Ulcer
Keywords: high ankle block; diabetes foot; wound healing; foot ulcer area; pulse perfusion index; hemodynamic parameters
MeSH Terms: conditions — Diabetic Foot | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAB group (Experimental): The superficial peroneal nerve, deep peroneal nerve, tibial nerve, gastrocnemius nerve, and saphenous nerve were sequentially blocked from one-third of the lower leg to the middle leg (about 15cm above the inner or outer ankle). 0.375% ropivacaine is used for the block and the total dose is 35ml. The ultrasound probe is placed vertical to the longitudinal axis of the body. On the lateral of tibia and fibula, 5ml of local anesthetic was injected to block the superficial peroneal nerve and 10ml for the deep peroneal nerve. On the posterior of the calf, 10ml of local anesthetic was injected to block the tibial nerve and 5ml for the sural nerve. On the inner side of the calf, 5ml of local anesthetic was injected to block the saphenous nerve.
  Interventions: Procedure: high ankle block
- GA group (Placebo Comparator): No nerve block, only general anesthesia with tracheal intubation.
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: high ankle block — The block position is in the middle and lower third of the calf, about 15cm above the inner or outer ankles. 0.375% ropivacaine is used for the block and the total dose is 35ml. The ultrasound probe is placed vertical to the longitudinal axis of the body. On the lateral of tibia and fibula, 5ml of local anesthetic was injected to block the superficial peroneal nerve and 10ml for the deep peroneal nerve. On the posterior of the calf, 10ml of local anesthetic was injected to block the tibial nerve and 5ml for the sural nerve. On the inner side of the calf, 5ml of local anesthetic was injected to block the saphenous nerve. The "water separation" technique is used and 2ml of physiological saline is injected before blocking to clarify the position of the needle tip and avoid nerve damage. 20 minutes after, the effect was measured using acupuncture by visual analogue scale (VAS) score. If the VAS score is less than 3, the block is considered successful and surgery is immediately performed.
  Arms: HAB group
Procedure: general anesthesia — intravenous injection of midazolam 0.03-0.05 mg/kg, etomidate 0.15-0.20 mg/kg, cisatracurium 0.15-0.20 mg/kg, and sufentanil 0.3-0.5 μg/kg. Intraoperative anesthesia maintenance using intravenous infusion of remifentanil 0.1-0.3 μg/kg·min, propofol 4-6 mg/kg·h, maintain bispectral index (BIS) value of 40-60, maintain intraoperative blood pressure and heart rate fluctuations within ± 20% of the baseline value, intermittently inject cisatracurium intravenously as needed. After the surgery, the patient was transferred to post-anaesthesia care unit (PACU). After regaining consciousness and regaining autonomous breathing, the tracheal catheter was removed and transferred to the ward when the indications for transfer were met.
  Arms: GA group

SUMMARY:
The goal of this clinical trial is to compare high ankle block and general anesthesia on wound recovery and ankle blood flow perfusion after diabetes foot surgery in diabetics. The main questions it aims to answer are:

* weather the high ankle block can fast wound recovery after the surgery
* weather the high ankle block can improve ankle blood flow perfusion after the surgery Participants will receive either high ankle block or general anesthesia during surgery. After the operation, foot ulcer area and pulse perfusion index will be measured on the postoperative day of 1 and 14; lower limb hemodynamic parameters will be measured by ultrasound on the postoperative days of 1, 7, and 14.

Researchers will compare high ankle block and general anesthesia to see if they have the different on the wound recovery and blood flow perfusion of the patients' foot.

DETAILED DESCRIPTION:
Inclusion criteria: refer to the 2019 World Guide for the Prevention and Treatment of diabetes Feet (DF), DF patients who meet the diagnostic criteria were Wagner's grade 2-4, good communication skills and ability to co-operate in completing various monitoring operations. Exclusion criteria: Skin infection at the puncture site; Concomitant severe cardiovascular and cerebrovascular diseases; Significant abnormalities in coagulation function; Mental abnormalities; Dementia and cognitive impairment. Patients were divided into a high ankle block group (HAB) and a general anesthesia group (GA) using a random number table method.

Regional procedures The patient fasted for 6 hours and stopped drinking for 2 hours before surgery without any preoperative medication. Routine hemodynamic and respiratory monitoring were performed upon entry. In the HAB group, the same senior anesthesiologist performed ultrasound-guided high ankle block on the affected side, with a local anesthetic formula of 0.25% ropivacaine 35ml. The superficial peroneal nerve, deep peroneal nerve, tibial nerve, gastrocnemius nerve, and saphenous nerve were sequentially blocked from one-third of the lower leg to the middle leg (about 15cm above the inner or outer ankle). The method is to place the long axis of the ultrasound probe perpendicular to the longitudinal axis of the body, and place it on the lateral front of the tibia and fibula of the calf. 5ml of local anesthetic is injected to block the superficial peroneal nerve and 10ml to block the deep peroneal nerve; 10ml of local anesthetic is injected to block the tibial nerve behind the calf; 5ml of local anesthetic into the posterior side of the calf to block the sural nerve; 5ml of local anesthetic on the inner side of the calf to block the saphenous nerve. The operation adopts the "water separation" technique, and 2ml of saline is injected before blocking each nerve to clarify the position of the needle tip and avoid nerve damage. 20 minutes after the completion of nerve block surgery, the visual analogue pain score (VAS) was measured using acupuncture, of which the areas innervated are the tibial nerve (posterior ankle and plantar), superficial and deep peroneal nerves (lateral calf and dorsal ankle), sural nerve (lateral calf and ankle), and saphenous nerve (medial calf and ankle). A VAS score of less than 4 indicates successful block, and surgery was performed immediately.

Patients in the GA group did not undergo nerve block and were given anesthesia induction and normal surgery after completing monitoring. Anesthesia induction: intravenous injection of midazolam 0.03-0.05 mg/kg, etomidate 0.15-0.20 mg/kg, cisatracurium 0.15-0.20 mg/kg, and sufentanil 0.3-0.5 μg/kg. Intraoperative anesthesia maintenance using intravenous infusion of remifentanil 0.1-0.3 μg/kg·min, propofol 4-6 mg/kg·h, maintain a BIS value of 40-60, maintain intraoperative blood pressure and heart rate fluctuations within ± 20% of the baseline value, intermittently inject cisatracurium intravenously as needed. After the surgery, the patient was transferred to PACU. After regaining consciousness and regaining autonomous breathing, the tracheal catheter was removed and transferred to the ward when the indications for transfer were met. Due to the weak postoperative pain stimulation after debridement surgery, neither group received additional postoperative pain pump analgesia. If the patient complained that the VAS score was greater than 4 points, the doctor would provide corresponding medication treatment according to the "three steps" of postoperative pain management.

Measurement of foot ulcer area and pulse perfusion index:

Follow up on the recovery of foot ulcers after surgery, take photos of the patient's ulcer surface using a mobile phone at T0, T7, and T14 time points, and calculate the foot ulcer area using NIH Image J (Version 1.46) software. The pulse oxygen saturation probe of the electrocardiogram monitor collects the T0, T7, and T14 pulse perfusion index (PI) of the first toe of the affected foot.

Measurement of arterial blood flow parameters:

After the nerve block is completed, the patient immediately returns to a supine position, with both legs exposed and in an outward rotation position (without touching each other). Use color Doppler ultrasound, take high-frequency linear array probe (frequency 10MHz), place the probe 3-5 cm above the ankle on the front side of the lower legs, look for the anterior tibial artery and the posterior tibial artery, first use the color two-dimensional mode to obtain the sagittal axis image of the artery, then use the pulse Doppler mode, the sampling volume is the size of the inner diameter l/3, place the middle of the blood vessel, and adjust the Doppler angle (the angle between the sound beam and the blood flow direction θ) Set at 60 °, record the arterial blood flow rate (FV), peak systolic velocity (PSV), end diastolic velocity (EDV), time mean velocity (TAmean), and time maximum mean velocity (TAmax) using automatic tracking method, and mark the position of the probe with a pen. The measurement time points were preoperative (T0), postoperative day 1 (T1), day 7 (T7), and day 14 (T14).

Measurement of skin temperature:

Using an infrared thermal imager (with a measurement resolution of up to 0.1 ℃), fixed on a lifting frame 30 cm away from the patient's ankle area skin, infrared thermal imaging images were collected and skin temperature was measured. The measurement areas were the thumb area, dorsum of foot area, and anterior tibia area. The measurement time points are T0, T1, T7, and T14, respectively. During the measurement period, instruct the patient not to move their legs.

After surgery, VAS was used to record the patient's pain scores on the first day (T1) and the second day (T2), with scores ranging from 0 to 10 indicating the degree of pain and the use of adjuvant analgesics.

ELIGIBILITY:
Inclusion Criteria:

* refer to the 2019 World Guide for the Prevention and Treatment of diabetes Feet (DF), DF patients who meet the diagnostic criteria were Wagner's grade 2-4, good communication skills and ability to co-operate in completing various monitoring operations.

Exclusion Criteria:

* Skin infection at the puncture site; Concomitant severe cardiovascular and cerebrovascular diseases; Significant abnormalities in coagulation function; Mental abnormalities; Dementia and cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
foot ulcer area | 1 day before operation, 1 day and 14 days after operation
  ulcer area of the diabetes Foot

SECONDARY OUTCOMES:
pulse perfusion index (PI) of the first toe | 1 day before operation, 1 day and 14 days after operation
  The pulse oxygen saturation probe of the electrocardiogram monitor collects the pulse perfusion index (PI) of the first toe of the affected foot.
arterial blood flow rate (FV) of anterior and posterior tibial arteries | 1 day before operation, 1 day, 7 days and 14 days after operation
  Use color Doppler ultrasound, take high-frequency linear array probe (frequency 10MHz), place the probe 3-5 cm above the ankle on the front side of the lower legs.
peak systolic velocity (PSV) of anterior and posterior tibial arteries | 1 day before operation, 1 day, 7 days and 14 days after operation
  Use color Doppler ultrasound, take high-frequency linear array probe (frequency 10MHz), place the probe 3-5 cm above the ankle on the front side of the lower legs.
end diastolic velocity (EDV) of anterior and posterior tibial arteries | 1 day before operation, 1 day, 7 days and 14 days after operation
  Use color Doppler ultrasound, take high-frequency linear array probe (frequency 10MHz), place the probe 3-5 cm above the ankle on the front side of the lower legs.
time mean velocity (TAmean) of anterior and posterior tibial arteries | 1 day before operation, 1 day, 7 days and 14 days after operation
  Use color Doppler ultrasound, take high-frequency linear array probe (frequency 10MHz), place the probe 3-5 cm above the ankle on the front side of the lower legs.
Toe and dorsum skin temperature | 1 day before operation, 1 day, 7 days and 14 days after operation
  infrared thermal imaging images were collected and skin temperature was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China